CLINICAL TRIAL: NCT00375310
Title: Phase I Study of Gemcitabine With Novel RAF Kinase-Vascular Endothelial Growth Factor Receptor Inhibitor Sorafenib (BAY 43-9006) and Radiotherapy in Patients With Locally Advanced Unresectable Pancreatic Adenocarcinoma
Brief Title: Phase I Study of Gemcitabine, Sorafenib and Radiotherapy in Patients With Unresectable Pancreatic Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Indiana University School of Medicine (Other)
Collaborators: Amgen (Industry)
Responsible Party: Sponsor
Organization: Indiana University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0607-09; IUCRO-0155
Record Dates: First submitted 2006-09-11; First posted 2006-09-12 (Estimated); Last update posted 2016-02-29 (Estimated); Status verified 2016-02

CONDITIONS: Pancreatic Cancer; Adenocarcinoma of the Pancreas
Keywords: Phase I; Pancreas Cancer; Chemo-radiotherapy
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Gemcitabine; Sorafenib; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Gemcitabine + Sorafenib & radiotherapy (Experimental): Induction: Gemcitabine with Sorafenib for 4 weeks (1 cycle). Chemo-radiotherapy: Gemcitabine with Sorafenib and Radiotherapy for 5 weeks. Sorafenib will be given in escalating dose cohorts.
  Sorafenib only: Sorafenib alone for 4 weeks. Consolidation: Gemcitabine with Sorafenib for 16 weeks (4 cycles). Maintenance: Sorafenib alone until disease progression.
  Interventions: Drug: Gemcitabine, Sorafenib; Procedure: Radiotherapy

INTERVENTIONS:
Drug: Gemcitabine, Sorafenib — Gemcitabine is given IV
  Sorafenib is given orally of varying doses:
  1. Sorafenib 200 mg po qd ( during combination therapy)
  2. Sorafenib 400 mg po qd ( during combination therapy)
  3. Sorafenib 400 mg po bid ( during combination therapy)
  Other Names: Gemzar ( gemcitabine); Sorafenib (BAY 43-9006)
Procedure: Radiotherapy — 1.8 Gy CTV daily for 5 weeks

SUMMARY:
The purpose of this study is to evaluate the safety and tolerability of the combined treatment of Sorafenib (BAY 43-9006) with Gemcitabine and radiotherapy in patients with localized unresectable pancreatic cancer.

DETAILED DESCRIPTION:
Pancreatic cancer treatment is hampered by its resistance to both chemo and radiotherapy. Gemcitabine-based chemoradiotherapy has become one of the standard therapies for localized unresectable pancreatic cancer, but with poor responses and survival rates of less than 12 months. Radiotherapy increases VEGF expression and activates the Ras/MEK/ERK pathway which may contribute to radioresistance, thus the addition of anti-angiogenic agents and/or Ras/ERK inhibitors could enhance radiation mediated cytotoxicity. Sorafenib is a novel dual-action Raf kinase and vascular endothelial growth factor receptors (VEGF-R2 and VEGF-R3) inhibitor targeting both angiogenic and Ras-Raf-1 signal transduction pathways. Based upon preliminary laboratory and clinical data Sorafenib holds promise for improving outcomes of therapy for patients with locally advanced unresectable pancreatic cancer.

Polymorphisms in genes involved in the angiogenesis pathway (VEGF, VEGF-R2, HIF-1 and eNOS) may contribute to the process of angiogenesis, tumor behavior, and may explain the heterogeneity in efficacy (and toxicity) of agents whose major mechanism of action is blocking angiogenesis33-37. Proteomic analysis may also contribute to identify patterns of response or resistance to therapies, and potentially predict outcomes.

Dynamic contrast enhanced (DCE)-MRI has been shown to be a useful pharmacodynamic marker of biological activity for anti-angiogenic agents38-40 and may also predict radiation therapy-induced vascular changes41. In vivo imaging of angiogenesis using DCE-MRI and the analysis of angiogenesis markers genetic polymorphisms may predict response and clinical benefit to therapy for unresectable pancreatic cancer patients. These biologic and pharmacodynamic endpoints will be analysed to correlate with the tumor activity seen.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically/pathologically confirmed locally advanced unresectable or borderline unresectable pancreatic cancer & no evidence of metastatic disease. Diagnosis of locally advanced unresectable pancreatic cancer is based on assessment by dual-phase CT scan and/or endoscopic ultrasound (EUS).
2. Age ≥ 18 years at time of consent
3. Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1
4. Measurable disease according to Response Evaluation Criteria in Solid Tumors (RECIST) & obtained by dual-phase CT scan within 14 days prior to being registered for protocol therapy.
5. Tumor size ≥ 2 cm on dual-phase computed tomography scan.
6. Adequate organ function documented within 14 days of registration as laboratory tests per protocol.
7. Patients with biliary obstruction must have percutaneous transhepatic drainage or endoscopic stent placement prior to starting study treatment
8. Women of childbearing potential must have a negative serum pregnancy test performed within 7 days prior to the start of treatment. Women of childbearing potential & men must agree to use adequate contraception (barrier method of birth control) prior to study entry & for the duration of study participation & for at least three months after the last administration of sorafenib.
9. Ability to understand & the willingness to sign a written informed consent. A signed informed consent & authorization for release of personal health information must be obtained prior to any study specific procedures.
10. Patients with a history of malignancy are eligible provided they have been curatively treated & demonstrate no evidence for recurrence of that cancer.

Exclusion Criteria:

1. Prior treatment with Gemcitabine within 6 months prior to registration.
2. Prior treatment with Sorafenib or other Ras or VEGF pathway inhibitors.
3. Prior radiation therapy to the upper abdomen
4. Evidence of metastatic disease
5. Clinical evidence of duodenal mucosal invasion by tumor (as documented by endoscopy or endoscopic ultrasound).
6. Minor surgical procedure (e.g. fine needle aspiration or needle biopsy) within 14 days of study registration.
7. Major surgical procedure, significant traumatic injury, or serious non-healing wound, ulcer or bone fracture within 21 days of study registration; investigator has to document adequate healing has occurred prior to study registration.
8. Any of the following within 6 months prior to study drug administration: severe/unstable angina (anginal symptoms at rest), new onset angina (began within the last 3 months) or myocardial infarction, congestive heart failure, cardiac ventricular arrhythmias requiring anti-arrhythmic therapy.
9. History of thrombotic or embolic events such as cerebrovascular accident or transient ischemic attack within the past 6 months. History of aneurysm or arteriovenous malformation.
10. Known human immunodeficiency virus (HIV) infection or chronic Hepatitis B or C.
11. Active clinically serious infection > Common Toxicity Criteria for Adverse Effects (CTCAE) grade 2.
12. Receipt of any investigational agent within 4 weeks of study registration.
13. Uncontrolled hypertension defined as systolic blood pressure > 150 mmHg or diastolic pressure > 90 mmHg, despite optimal medical management.
14. Pulmonary hemorrhage/bleeding event > CTCAE Grade 2 within 4 weeks of study registration
15. Any other hemorrhage/bleeding event > CTCAE Grade 3 within 4 weeks of study registration
16. Evidence or history of bleeding diathesis or coagulopathy.
17. Chronic, daily treatment with aspirin or other nonsteroidal anti-inflammatory medications.
18. Use of St. John's Wort, rifampin (rifampicin), ketoconazole, itraconazole, ritonavir or grapefruit juice.
19. Known or suspected allergy to Sorafenib or any agent given in the course of this trial.
20. Any condition that impairs patient's ability to swallow whole pills.
21. Any malabsorption problem.
22. Other severe, acute or chronic medical or psychiatric condition, or laboratory abnormality that may increase the risk associated with study participation or study drug administration, or may interfere with the interpretation of study results & in the judgment of the investigator would make the patient inappropriate for entry into this study.
23. History of collagen vascular disease.
24. Any contraindication to undergo magnetic resonance imaging

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2006-09; Primary Completion 2010-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
To evaluate the safety and tolerability of the combined treatment with Gemcitabine with Sorafenib and radiotherapy in patients with localized unresectable pancreatic cancer. | completion of study

SECONDARY OUTCOMES:
To evaluate the response rate (CR + PR), clinical benefit (CR + PR + SD) and tumor shrinkage (CR + PR + SD that shrinks) of Gemcitabine with Sorafenib and radiotherapy | completion of study
To evaluate time to disease progression and overall survival. | completion of study
To evaluate pharmacodynamic changes in tumor vascular parameters (e.g blood flow, blood volume, time to peak in ROC -receiver operator characteristics curve) by DCE-MRI and correlate with outcomes. | completion of study
To evaluate biologic markers such as VEGF, eNOS and HIF1-alpha, VEGF-R2 genetic polymorphisms and serum proteomics, and correlate with outcomes. | completion of study
To evaluate resectability rates of tumors after treatment. | completion of treatment
To evaluate the maximum tolerated dose (MTD) for Sorafenib during Chemo-radiation. | completion of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Romnee Clark, MD, Principal Investigator — IU Simon Cancer Center
Locations (1):
- Indiana University Simon Cancer Center, Indianapolis, Indiana, United States